CLINICAL TRIAL: NCT04401501
Title: Short- and Mid-Term Effects of Manual Therapy on the Upper Cervical Spine Combined With Exercise vs Isolated Exercise in Patients With Cervicogenic Headache. A Randomized Controlled Trial.
Brief Title: Effects of Manual Therapy on the Upper Cervical Spine Combined With Exercise vs Isolated Exercise in Patients With Cervicogenic Headache.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Jacobo Rodríguez-Sanz, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N14/2020
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2020-05

CONDITIONS: Cervicogenic Headache; Headache
Keywords: Cervicogenic headache; exercise; manual therapy; upper cervical spine
MeSH Terms: conditions — Post-Traumatic Headache; Headache; Motor Activity | interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy + Exercise Group (Experimental): Combination of manual therapy and exercises for cervicogenic headache
  Interventions: Other: Manual Therapy and Exercises
- Exercise Group (Active Comparator): Only exercises for cervicogenic headache
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Manual Therapy and Exercises — Combination of physiotherapy (manual therapy) techniques and exercises for cervicogenic headache
  Arms: Manual Therapy + Exercise Group
Other: Exercise — Exercises for cervicogenic headache
  Arms: Exercise Group

SUMMARY:
Cervicogenic headache is defined as unilateral headache associated with neck pain. Effect of manual translatoric therapy of the upper cervical spine associated with cervical exercises in these patients is currently unknown. Our aim was to determine if adding manual therapy to an exercise and home-exercise program improved effects on symptoms and function in short- and mid-term in patients with cervicogenic headache.

A randomized controlled study will be conducted with 40 subjects with cervicogenic headache. Each group will receive four 20-minute sessions weekly and a home-exercise program. Upper cervical flexion, flexion-rotation test, Impact Headache Test-6 (HIT-6), headache intensity, craniocervical flexion test, pain pressure thresholds and Global Rating of Change (GROC)-Scale will be assessed at end of the intervention, at 3- and at 6-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cervicogenic headache according to Sjaastad et al. Subjects will have to fulfill both parts I and III of the major criteria for diagnosis (pain aggravated by neck movement, sustained position or external pressure, restricted cervical range of motion, and unilateral pain starting in the neck and radiating to the frontotemporal region)
* Hypomobility in one or more segments of C0-1, C1-2, C2-3 through manual evaluation.
* A positive result in the flexion-rotation test.
* A failure to pass stage 2 (24 mmHg) of the craniocervical flexion test.
* Be at least 18 years old.
* Have signed the informed consent.

Exclusion Criteria:

* Contraindications for manual therapy or exercise.
* Participation in exercise or manual therapy programs in the last three months.
* Inability to maintain supine position.
* The use of pacemakers (the magnets in the CROM device could alter their signal).
* Inability to perform the flexion-rotation test.
* Language difficulties.
* Pending litigation or lawsuits.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Headache Intensity (HIT-6) | Change between baseline and post intervention (1 month), after 3 months and after 6 months
  Test-6 questionnaire (HIT-6) will be used to describe the degree of pain and disability caused by the headache, with a reliability higher than 0.70. The results are classified into four categories that score daily life impact of headache (little or none, some, substantial and severe.
Flexion-rotation test | Change between baseline and post intervention (1 month), after 3 months and after 6 months
  This test is used to see the amount of movement of the upper cervical spine and is the test most used in the literature. It is positive when there is a decrease of 10 degrees or more in the cervical rotation with maximum flexion, in a sense with respect to the contralateral or presents hypomobility of segment C1 with a mobility less than 32º

SECONDARY OUTCOMES:
Upper cervical flexion range of motion | Change between baseline and post intervention (1 month), after 3 months and after 6 months
  Active flexion of the upper cervical spine will be measured in standing position using a CROM device
Headache Intensity | Change between baseline and post intervention (1 month), after 3 months and after 6 months
  Headache intensity will be assessed on a visual analogue scale from 0 to 10 cm.
Craniocervical flexion test | Change between baseline and post intervention (1 month), after 3 months and after 6 months
  This test will be used to measure the strength of the deep flexor muscles. The activation and resistance of the deep flexor muscles will be evaluated in five progressive pressure increases of 2 mmHg up to a maximum of 30 mmHg. The patient will pass to the next level after reaching one certain level three times.
Pain Pressure Thresholds | Change between baseline and post intervention (1 month), after 3 months and after 6 months
  Pain pressure thresholds will be measured using a digital algometer (Somedic AB Farsta, Somedic SenseLab AB, Sweden) with a round surface area of 1 cm2. Pressure will be applied at a rate of 1 kg/cm2/s, perpendicular to the skin. Pressure pain thresholds will be assessed over six points bilaterally with the subject in supine position: suboccipital region, C2-3, C5-6, elevator of scapula, trapezius and first metacarpal joint.
Global Raiting of Scale (GROC-Scale) | Change between baseline and post intervention (1 month), after 3 months and after 6 months
  GROC-Scale will be used to measure the personal evolution that the patient had experienced. This scale is considered to be an efficient way to score patients' perceived clinical change and test-reliability has shown to be excellent (ICC=0.90).
Adherence to self-treatment scale | Change between baseline and post intervention (1 month), after 3 months and after 6 months
  This scale will be used in order to measure the adherence to self-treatment at home. Patients will be asked to choose between the following answers: "I have done the exercises every day"; "I have performed the exercises 4-6 days a week"; "I have performed the exercises 1-3 days a week"; "I have performed the exercises less than 1 day a week"; or "I have not performed them".

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Zaragoza, Zaragoza, Spain